CLINICAL TRIAL: NCT03828578
Title: Comparison of AIRVO High Flow Oxygen Therapy With Standard Care for Prevention of Post-operative Pulmonary Complications After Major Head and Neck Surgery Involving Insertion of a Tracheostomy - A Proof of Concept Study
Brief Title: Comparison of AIRVO High Flow Oxygen Therapy With Standard Care for Prevention of PPCs After Major H&N Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Principal Investigator, Paul Twose, Physiotherapist, Cardiff and Vale University Health Board
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 223048
Record Dates: First submitted 2019-01-19; First posted 2019-02-04 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow oxygen therapy (Experimental): Patients allocated to the intervention group will receive high flow oxygen therapy via the tracheostomy tube from cessation of mechanical ventilation. The HFOT will provide oxygen therapy at a flow rate of 50-60 litres per minute at a FiO2 titrated by the bedside clinician to maintain a peripheral oxygen saturation of 95% of more (unless otherwise clinically indicated and documented by an appropriate consultant).
  Once transferred to the ward patients will continue to receive HFOT 24 hours per day at a rate of 50-60 litres per minute at a maximum oxygen concentration of 40% to achieve oxygen saturations 95% and above (unless otherwise documented).
  Patients may be disconnected from the HFOT for short periods for toileting, mobilising etc. Tracheostomy weaning will continue as per standard practice with an aim of cuff deflation followed by decannulation once clinically appropriate. systems. Following decannulation patients will resort to standard oxygen therapy as needed.
  Interventions: Procedure: High flow oxygen therapy
- Standard Care (No Intervention): Patients randomised to the standard care study arm will receive routine post-operative care as currently performed within the host organisation. Following cessation of mechanical ventilation, oxygen therapy will be delivered using equipment and rates appropriate to the clinical picture. On transfer to the ward patients will continue with existing methods of oxygen therapy and will be weaned from these accordingly. Patients will continue to use heat moisture exchanges (e.g. Swedish nose or Buchannan protectors) as clinically indicated, as well as having saline nebulisers prescribed and administered as per standard. Tracheostomy weaning will continue in accordance with current practice. Data on all of the applied procedures will be recorded.

INTERVENTIONS:
Procedure: High flow oxygen therapy — High flow oxygen therapy delivered via Airvo2
  Arms: High flow oxygen therapy

SUMMARY:
Patients undergoing major head and neck surgery often develop breathing difficulties as a result of build up of sputum and difficulty taking deep breaths. Often as part of the surgery patients may also require a tracheotomy tube (a temporary tube placed into their airway) which is removed around 5-7 days after the operation. The presence of this tracheostomy tube increases the patient's risk of developing breathing problems, especially difficulty clearing sputum and reduced lung volumes. To reduce the risk of developing these problems, different forms of oxygen therapy and humidification are used. This normally involves using oxygen masks, nebulisers and other medications to help loosen the sputum and maintain blood oxygen levels. Another method of giving oxygen and humidification is through the use of AIRVO, which delivers the air / oxygen to the patient at higher rates as well as warming and humidifying the air.

The aim of this study is to compare the AIRVO system to standard care in a small sample of patients (20 patients) undergoing major head and neck surgery involving insertion of a tracheostomy tube.

The study will compare rates of breathing complications (e.g. pneumonia, reduced lung volume) as well as comparing the time to remove the tracheostomy tube and the time the patient is required to stay in hospital. These results will then be used to develop a larger funded study.

DETAILED DESCRIPTION:
Major head and neck surgery involving micro-vascular reconstructions are prolonged procedures with considerable post operative risk. Not only do patients have prolonged time in theatre, the surgery involves two distinct surgical sites (head & neck site and peripheral flap donor site), and requires the patient to be admitted to a high care area for overnight sedation and ventilation. This combined with the presence of significant co-morbidities such as hypertension, cardiomyopathy and respiratory disease, place the patient at significant risk of post-operative complications. A recent prospective cohort study reported complication rates in nearly 65% of cases, of which 29% were of pulmonary origin. Furthermore, of these, 14 patients required treatment in the intensive care or high dependency. Interestingly, and in contrast to other research3, neither pre-operative smoking nor the presence of pre-existing lung disease predicted pulmonary complications.

The risks of post-operative pulmonary complications (PPCs) seem to be further increased in those patients requiring a tracheostomy. This tracheostomy is required to facilitate access to the tumour location and to provide post-operative airway protection in the presence of significant swelling or oedema. The risks of tracheostomy are well known4. Patients are prone to increased rates of infection, poor sputum clearance and inadequate humidification. These complications lead to prolonged admissions, delays in tracheostomy weaning and considerable healthcare related costs. To overcome these issues national guidance documents have identified the need to provide adequate humidification to prevent mucus plugging, as well as the provision of increased nursing care for stoma site cleaning and inner tube care. Historically, humidification has been provided by heated systems however due to perceived increased infection risk this has fallen out of favour and now passive humidification systems such as heat moisture exchangers have become more popular.

Clearly, the combination of the risks of major head and neck surgery and those of a tracheostomy, place the patient at significant risk. As such it is essential to develop new post-operative management protocols to reduce the occurrence of post-operative complications.

AIRVOTM (a form of non-invasive high flow oxygen therapy, HFOT), which delivers high flow heated and humidified oxygen and air via a tracheostomy tube at a prescribed fraction of inspired oxygen and a maximum flow of 60 L/min, is an attractive alternative to conventional oxygen therapy. Previous studies have shown that HFOT therapy generates a flow-dependent positive airway pressure and improves oxygenation by increasing end-expiratory lung volume, thus suggesting a possible alveolar recruitment associated with high-flow therapy. Although widely used in other clinical areas including patients with tracheostomy tubes, HFOT delivered in the AIRVOTM system has yet to be evaluated in the Head and Neck surgery population.

This study aims to compare the effects of application of HFOT(delivered via AIRVOTM) therapy and conventional oxygen and humidification administration after major head and neck surgery involving insertion of a tracheostomy tube on postoperative pulmonary complications. The study will also compare post-operative length of stay, time to tracheostomy tube cuff deflation, tracheostomy tube decannulation, antibiotic use and post-operative physiotherapy requirements.

The results of this proof of concept study will be used to further develop local protocols and to inform a grant funded multi-centre trial.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing head and neck surgery with microvascular reconstruction and involving insertion of a tracheostomy

Exclusion Criteria:

* Under 18 years old
* Lack of consent
* Consultant request

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants diagnosed with post-operative Pulmonary Complications | Up to 48hours post tracheostomy decannulation

SECONDARY OUTCOMES:
Time to decannulation | Up to 4 weeks
  Measured in days
Hospital length of stay | Up to 4 weeks
  Measured in days
Amount of physiotherapy intervention recieved by each participant | Up to 4 weeks
  Measured in minutes
Feasability of recruitment, randomisation, delivery of intervention, and completion of outcome measures | Up to 4 weeks
  Measured in percentages

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiff and Vale University Health Board, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No